CLINICAL TRIAL: NCT06650956
Title: Integrated Service Delivery to Improve Adolescent Health and HPV Vaccination in Lao PDR: a Quasi-Experimental Mixed-Methods Study
Brief Title: Integration to Improve Adolescent Health and HPV Vaccination in Laos
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Health Poverty Action (Other)
Collaborators: Gavi, The Vaccine Alliance (Other); University of Health Sciences Laos (Unknown)
Responsible Party: Principal Investigator, Dr. Thet Lynn, Program Development and Quality Manager - Asia Region, Health Poverty Action
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 833/REC; Research Ethics Committee (Other: University of Health Sciences Laos)
Record Dates: First submitted 2024-10-09; First posted 2024-10-21 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Healthy; Adolescents; Integrated, Community-Health Systems; HPV Vaccines; Sexual and Reproductive Health; Knowledge; Attitude; Health Workers
Keywords: hpv vaccination; adolescent health; integration; lao pdr; cervical cancer prevention; sexual and reproductive health
MeSH Terms: conditions — Coitus; Behavior | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Intervention Model Description: The study population includes girls aged 10-13 years for HPV vaccination and boys and girls aged 10-13 years for other adolescent health services. The intervention district will receive an integrated service package comprising HPV vaccination and adolescent health services delivered through school-based, facility-based, and outreach approaches. The comparison district will continue with its standard HPV vaccination and routine adolescent health service delivery. The intervention will be for 7 months from 2024 November to 2025 May.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention district (Experimental): The intervention provides HPV vaccinations to girls aged 10-13 and sexual and reproductive health (SRH) services to boys and girls aged 10-13 through three service delivery touch points: schools, health facilities, and community outreach. The vaccine in the intervention is a single dose of recombinant Human Papilloma virus quadrivalent types, 6, 11, 16, and 18. Schools will provide vaccinations and comprehensive sexuality education (CSE) sessions. Health facilities offer vaccinations and SRH education service. Community outreach delivers the integrated package to out-of-school girls and boys.
  Interventions: Other: Integrated HPV and SRH Service Package; Biological: Human Papillomavirus Quadrivalent (Types 6, 11, 16, and 18) Vaccine, Recombinant
- Comparison District (Active Comparator): Standard HPV Vaccination (Comparison District) - In the comparison district, routine HPV vaccination services will be provided to girls aged 10-13 years. The vaccine is a single dose of recombinant Human Papilloma virus quadrivalent types, 6, 11, 16, and 18.; A school-based vaccination campaign will be conducted in 2024 November to promote and administer the HPV vaccine. Additionally, the vaccine will be available at health facilities starting in the same month. Outreach activities will also be conducted to ensure access to the vaccine for hard-to-reach populations and out-of-school girls. - Unlike the intervention district, there will be no additional training for nor service by healthcare providers on comprehensive sexuality education (CSE) or other sexual and reproductive health (SRH) services, and there will be no dedicated community outreach sessions on SRH topics.
  Interventions: Biological: Human Papillomavirus Quadrivalent (Types 6, 11, 16, and 18) Vaccine, Recombinant

INTERVENTIONS:
Other: Integrated HPV and SRH Service Package — 1. Integrated Service Package combines HPV vaccination with sexual and reproductive health (SRH) education. The vaccine in the intervention package is a single dose of recombinant Human Papilloma virus quadrivalent types, 6, 11, 16, and 18.;
  2. The package will be delivered through multiple touch-points such as school-based programs, health facility services, and community outreach. i) In school, the intervention incorporates Comprehensive Sexuality Education, empowering boys and girls with knowledge about their bodies, health, and rights. This goes beyond simply providing information about HPV and vaccination. ii) At health facilities, the intervention package will also be delivered in adolescent-friendly ways, ensuring that boys and girls feel comfortable accessing SRH information. iii) Since not all boys and girls attend school, the intervention includes community outreach that ensures wider reach and accessibility for adolescents aged 10-13, including those not enrolled in school.
  Arms: Intervention district
Biological: Human Papillomavirus Quadrivalent (Types 6, 11, 16, and 18) Vaccine, Recombinant — The vaccine itself is not the intervention of interest as this is delivered in both intervention and comparison arms. The vaccine is a single dose of recombinant Human Papilloma Virus Quadrivalent (Types 6, 11, 16, and 18). The administration of the vaccine is an intramuscular injection of 0.5 mili liter of suspension form.
  Other Names: Gardasil

SUMMARY:
The goal of this study is to find out if adding HPV vaccination to adolescent health services works to increase HPV vaccine uptake in 10-13-year-old girls in Laos. The study will also look at the effects of adding HPV vaccination on the use of other health services in 10-13-year-old boys and girls.

The main questions the study aims to answer are:

1. Does adding HPV vaccination to adolescent health services increase HPV vaccine uptake in girls aged 10-13 years compared to girls who only receive standard HPV vaccination services?
2. Does adding HPV vaccination to adolescent health services increase the use of other health services in 10-13-year-old adolescent boys and girls compared to adolescents who only receive standard HPV vaccination services?
3. What are the barriers and facilitators to using the combined intervention in Laos?
4. What are the opinions of adolescents, caregivers, healthcare providers, and other stakeholders on the combined intervention?
5. How much does it cost and how well it works to combine HPV vaccination with adolescent health services, as opposed to providing HPV vaccination alone?

Researchers will compare a combined intervention to standard HPV vaccination services to see if the combined intervention works to increase HPV vaccination uptake and the use of other health services. The combined intervention includes HPV vaccination given at schools, health facilities, and through community outreach. It also includes education on sexual and reproductive health, counseling, and other health services. Participants in the combined intervention group will:

1. Receive the HPV vaccine at school or at a health facility.
2. Take part in group discussions about sexual and reproductive health.
3. Take part in individual counseling sessions.
4. Use other health services as needed.

Participants in the comparison group will receive standard HPV vaccination services, including:

• HPV vaccination given at schools, health facilities, and through community outreach.

DETAILED DESCRIPTION:
Objectives: The overall objective of the study is to determine how integrating HPV vaccination services with adolescent health services could increase HPV vaccine coverage equitably and sustainability, as well as contribute to selected adolescent health outcomes in Lao.

Specific Objectives (SO):

1. To determine the extent to which the integration of HPV vaccination with adolescent health services increases HPV vaccine uptake among 10-13-year-old girls in the intervention district compared to the comparison district over 9 months.
2. To assess the impact of the integrated intervention on adolescents' knowledge, attitudes, and practices related to sexual and reproductive health and rights (SRHR) among 10-13-year-old boys and girls, as well as their utilization of other adolescent health services.
3. To identify barriers and facilitators to implementing the integrated intervention in the Laotian context, including its impact on healthcare providers' workload and capacity.
4. To explore the perceptions of adolescents, caregivers, healthcare providers, and other stakeholders regarding integrated intervention, including its perceived benefits and challenges.
5. To determine the costs and effects of integrating HPV vaccination with adolescent health services compared to delivering HPV vaccination alone and assess the cost-effectiveness of the integrated intervention in the Laotian context. [A separate protocol will be developed for full methodology to determine the cost and effects.]

Research Questions:

SO-1: 1.1) What is the difference-in-differences (DID) of change in the HPV vaccine uptake in the 10-13-year-old girls' population between the intervention and comparison districts over 9 months? 1.2) What factors contribute to the differences - if any - in HPV vaccine uptake as such between the intervention and comparison districts?;

SO-2: 2.1) How does the integrated intervention affect 10-13-year-old adolescents' knowledge, and attitudes related to SRHR in the intervention district compared to the comparison district over 9 months?, 2.2) What changes in the utilization of adolescent health services among 10-13-year-olds are observed in the intervention district compared to the comparison district?;

SO-3: 3.1) What are the main barriers and facilitators to implementing the integrated intervention in the Lao context?, 3.2 How does the integrated intervention impact healthcare providers' workload and capacity in the intervention district?;

SO-4: 4.1) What are the perceptions of adolescents, caregivers, healthcare providers, educators and other key stakeholders regarding the benefits and challenges of the integrated intervention?, 4.2) How do the perceived benefits and challenges of the integrated intervention vary among different stakeholder groups?;

SO-5: 5.1) What are the costs and effects of integrating HPV vaccination with adolescent health services compared to delivering HPV vaccination alone?, 5.2) How does the cost-effectiveness of the integrated intervention compare to that of delivering HPV vaccination alone in the Lao context?

ELIGIBILITY:
Inclusion Criteria:

* Female aged 10-13 years for HPV vaccination and SRH education
* Male aged 10-13 years for SRH education
* 10-13-year-old male and female students in randomly selected schools with at least 100 students in target classes (year-5 primary, year-1, 2 and 3 secondary)
* 10-13-year-old males and females who are out-of-school and living in 2 remote villages each from four randomly selected health centers located around the selected schools

Exclusion Criteria:

* males and females younger than 10 years or older than 13 years

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 700 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Difference-in-differences of HPV Vaccination Rates | Baseline: Assessment at the start of the study (Month 0). Mid-Intervention: Assessment 3 months after the intervention begins (Month 3). End-of-Intervention: Assessment 7 months after the intervention begins (Month 7)
  Difference-in-differences (DID) of the HPV vaccination rates in the 10-13-year-old girls' population between the intervention and comparison districts over 7 months

SECONDARY OUTCOMES:
Change in Scores of Knowledge and Attitude (KA) related to Sexual and Reproductive Health among adolescents | Baseline: Assessment at the start of the study (Month 0). Mid-Intervention: Assessment 3 months after the intervention begins (Month 3). End-of-Intervention: Assessment 7 months after the intervention begins (Month 7)
  This will measure change in scores of 10-13-year-old adolescents' knowledge, and attitude (KA) questionnaire related to SRH in the intervention district compared to the comparison district over 7 months
  The knowledge and attitude (KA) questionnaire is a structured assessment tool designed to measure participants' knowledge, attitudes, and practices related to sexual and reproductive health. It covers various aspects of SRH, including:
  1. Knowledge of HPV, cervical cancer, and prevention methods, and
  2. Attitudes towards HPV vaccination and sexual health.
  The questionnaire employs a variety of question formats, including multiple-choice, true/false, and Likert scales.
  Knowledge: 40 items (0-40 score range). Higher scores mean better knowledge. Attitude: 20 items (20-100 score range). Higher scores generally indicate more positive attitudes, but some items need reverse-scoring.
  Higher total scores mean better knowledge and more positive attitudes.
Themes on Barriers to Integrated HPV Vaccination and Adolescent Health Services in Lao PDR | End-of-Intervention: Assessment 7 months after the intervention begins (Month 7)
  Focus group discussions (FGDs) will be used to explore the consolidated themes on barriers encountered during the intervention.
  FGDs: Focus group discussions (FGDs) will be conducted with healthcare providers, educators, community leaders, caregivers and policymakers to gather diverse perspectives on the barriers to implementing the integrated intervention.
  The information from different groups will be aggregated by identifying common themes and patterns across the different groups, and these consolidated themes on barriers will be reported as the key findings for this outcome measure.
Themes on Healthcare Providers' Workload in Delivering Integrated HPV Vaccination and Adolescent Health Services | End-of-Intervention: Assessment 7 months after the intervention begins (Month 7).
  FGDs will be conducted to explore the themes on healthcare providers' workload for delivering the integrated intervention.
  FGDs: Focus group discussions (FGDs) will be conducted with healthcare providers to gather diverse perspectives on how the integrated intervention has affected their workload. The discussions will explore the changes in workload associated with the integration of HPV vaccination and SRH services, the adequacy of resources and training, and the overall impact on service delivery.
Themes on Perceptions of Stakeholders on Integrated HPV Vaccination and Adolescent Health Services | End-of-Intervention: Assessment 7 months after the intervention begins (Month 7).
  This outcome measure will assess consolidated thematic perceptions among various stakeholders regarding the integrated intervention, including its perceived benefits, challenges, acceptability and suggestions for improvement. Information will be gathered through IDIs and analyzed to identify key themes and areas of consensus and disagreement among stakeholders.
  IDIs: In-depth interviews (IDIs) will be conducted with a range of stakeholders, including:
  1. Adolescents who have participated in the intervention
  2. Caregivers of adolescents
  3. Healthcare providers involved in delivering the integrated services
  4. Educators who have participated in CSE
  5. Policymakers involved in adolescent health and vaccination programs
  The information gathered from different stakeholders will be aggregated by identifying common themes and patterns across the different groups, and these consolidated thematic perceptions will be reported as the key findings for this outcome measure.
Cost per unit delivery of integrated intervention package to the adolescents | End-of-Intervention: Assessment 7 months after the intervention begins (Month 7).
  To get the cost per unit delivery of integrated intervention package, the total cost will be divided by the total number of adolescents reached.
  The total cost of the intervention will be calculated by summing up all the costs collected across different cost components. All relevant cost components will be identified, including direct costs (i.e., vaccine procurement, personnel, training, materials) and indirect costs (i.e., overhead and transportation). The total number of adolescents reached will be calculated by the number of adolescents reached through different delivery channels (school-based, facility-based and community outreach).
Themes on Facilitators to Integrated HPV Vaccination and Adolescent Health Services in Lao PDR | End-of-Intervention: Assessment 7 months after the intervention begins (Month 7)
  Focus group discussions (FGDs) will be used to explore the consolidated themes on facilitators encountered during the intervention.
  FGDs: Focus group discussions (FGDs) will be conducted with healthcare providers, educators, community leaders, caregivers and policymakers to gather diverse perspectives on the facilitators to implementing the integrated intervention.
  The information gathered from different groups will be aggregated by identifying common themes and patterns across the different groups, and these consolidated thematic facilitators will be reported as the key findings for this outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Thet Lynn, MD, MMedSc Global Health, Principal Investigator — Health Poverty Action; Vanphanom Sychareun, MD, PhD, Principal Investigator — University of Health Sciences Laos
Locations (1):
- Sing District, Luang Namtha Province, Muang Sing, Province, Laos

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: October, 2025 - Jun,2026

REFERENCES:
- [Background] Markowitz LE, Tsu V, Deeks SL, Cubie H, Wang SA, Vicari AS, Brotherton JM. Human papillomavirus vaccine introduction--the first five years. Vaccine. 2012 Nov 20;30 Suppl 5:F139-48. doi: 10.1016/j.vaccine.2012.05.039. PMID 23199957
- [Background] Engel D, Afeli ADJ, Morgan C, Zeck W, Ross DA, Vyankandondera J, Bloem P, Adjeoda KR. Promoting adolescent health through integrated human papillomavirus vaccination programs: The experience of Togo. Vaccine. 2022 Mar 31;40 Suppl 1:A100-A106. doi: 10.1016/j.vaccine.2021.11.021. Epub 2021 Nov 26. PMID 34844819
- [Background] Vongxay V, Albers F, Thongmixay S, Thongsombath M, Broerse JEW, Sychareun V, Essink DR. Sexual and reproductive health literacy of school adolescents in Lao PDR. PLoS One. 2019 Jan 16;14(1):e0209675. doi: 10.1371/journal.pone.0209675. eCollection 2019. PMID 30650100
- [Background] Aryal A, Clarke-Deelder E, Phommalangsy S, Kounnavong S, Fink G. Health system inequities in Lao People's Democratic Republic: Evidence from a nationally representative phone survey. Trop Med Int Health. 2024 Jun;29(6):518-525. doi: 10.1111/tmi.13997. Epub 2024 Apr 30. PMID 38685885
- [Background] Starrs AM, Ezeh AC, Barker G, Basu A, Bertrand JT, Blum R, Coll-Seck AM, Grover A, Laski L, Roa M, Sathar ZA, Say L, Serour GI, Singh S, Stenberg K, Temmerman M, Biddlecom A, Popinchalk A, Summers C, Ashford LS. Accelerate progress-sexual and reproductive health and rights for all: report of the Guttmacher-Lancet Commission. Lancet. 2018 Jun 30;391(10140):2642-2692. doi: 10.1016/S0140-6736(18)30293-9. Epub 2018 May 9. No abstract available. PMID 29753597
- See also: United Nations, Department of Economic and Social Affairs, Population Division. World Population Prospects: The 2022 Revision — https://population.un.org/wpp/
- See also: GBD Compare. Seattle, WA: IHME, University of Washington: Institute for Health Metrics and Evaluation (IHME).; 2023 — http://ihmeuw.org/6h6b
- See also: Bruni L, Albero G, Serrano B, Mena M, Collado J, Gómez D, et al. Human Papillomavirus and Related Diseases in Laos. Summary Report 2023. ICO/IARC Information Centre on HPV and Cancer (HPV Information Centre) — https://hpvcentre.net/statistics/reports/LAO.pdf?t=1718017698721
- See also: Human papillomavirus and related cancers in Laos. Summary report 2010. WHO/ICO Information Centre on HPV and Cervical Cancer (HPV Information Centre) — http://www.hpvcentre.net/
- See also: Global strategy to accelerate the elimination of cervical cancer as a public health problem — https://iris.who.int/bitstream/handle/10665/336583/9789240014107-eng.pdf?sequence=1
- See also: Human papillomavirus vaccines: WHO position paper (2022 update). Weekly Epidemiological Record, 2022, vol 97, 50. 2022 Dec 16;97(50):645-72 — https://iris.who.int/bitstream/handle/10665/365350/WER9750-eng-fre.pdf?sequence=1